CLINICAL TRIAL: NCT02711046
Title: Evaluation of Change in Mouth Opening in Oral Submucous Fibrosis Patients After Surgical Excision of Fibrous Bands Along With Bilateral Coronoidotomy and Surgical Defect Coverage by Single Stage Extended Nasolabial Flap
Brief Title: Use of Single Staged Nasolabial Flap in Oral Submucous Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College of Dentistry, Indore (Other)
Responsible Party: Principal Investigator, Dr. Faisal Idrees, Dr., Government College of Dentistry, Indore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDCORALSURGERY
Record Dates: First submitted 2016-02-16; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Oral Submucous Fibrosis
MeSH Terms: conditions — Oral Submucous Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single stage nasolabial flap (Experimental): single staged nasolabial flap as an interpositional material after surgical resection of fibrous band in oral submucous fibrosis
  Interventions: Procedure: single stage nasolabial flap

INTERVENTIONS:
Procedure: single stage nasolabial flap — The versatility of this flap has been attributed to the fact that there is often abundant non-hair-bearing skin in this well-vascularized region. The facial and infraorbital arteries are frequently cited in anatomic descriptions of the nasolabial flap. The venous drainage is believed to be via the angular and facial veins.

SUMMARY:
Long standing oral submucous fibrosis(OSMF) is associated with involvement

of the oral submucosa and the muscles of mastication leading to difficulty in mouth

opening. Various surgical modalities are mentioned for release but each has its own limitations.The aim of the study was to evaluate the change in mouth opening in patients of OSMF after excision of fibrous bands followed by coronoidotomy and surgical defect coverage by single stage nasolabial flap.

DETAILED DESCRIPTION:
The world of medical science is replete with a plethora of conditions both physiological and pathological which exhibit manifold symptoms, some of which man has conquered while against others, he is still waging a relentless battle. In this fast changing world of stress and cut throat competition, we humans often resort ourselves to tension relieving habits like alcoholism, smoking, tobacco or betel nut chewing. Apart from the very severe systemic consequences of these habits, oral cavity is also very adversely affected. Of all the unique oral afflictions that these habits have on oral cavity of betel quid chewers, Oral Submucous Fibrosis (OSMF) holds a pivotal position.

OSMF is a distressing condition in which due to limited opening of the oral cavity, the patient is neither able to consume a normal diet nor maintain proper oral hygiene. OSMF mostly occurs in Asian countries, including India ,China, Pakistan, Sri Lanka and Bangladesh, where chewing betel quid (areca nut , tobacco, slaked lime, or other species) is very popular & accepted as form of tradition in most part of these countries. It is observed that irritants like betel nuts, tobacco etc. if kept for longer period around the cheek and swallowed gradually may play a major part in the causation of the disease.

In India, the first mention of this disease in literature dates back to time of 'Sushruta' as 'Vidari'. However in modern literature 'Schwartz' in 1952 first described it as "Atrophica idiopathica mucosa oris".

Oral submucous fibrosis is "an insidious, chronic disease affecting any part of the oral cavity and sometimes the pharynx. Although occasionally preceded by and/or associated with vesicle formation, it is always associated with a juxta-epithelial inflammatory reaction followed by a fibroelastic change of the lamina propria, with epithelial atrophy leading to stiffness of the oral mucosa causing trismus and inability to eat" Usually in this disease patient has no disabling symptoms in the early phase, but as it progress it causes burning sensation, difficulty in eating and opening of mouth, that forces patients to report a clinician with these distressing symptoms. Sharp (1956) has described submucous fibrosis along with epithelial hyperplasia and mucosal atrophy as a characteristic feature of abnormal-precancerous oral epithelium and of tissue adjacent to frank oral cancer. OSMF can transform into oral cancer, and particularly squamous-cell carcinoma, at a rate in the range of 7% to 13%.

OSMF can occur in any decade of life but is commonly seen in 2nd -4th decade of life. Various studies have suggested multifactorial origin of the disease with high incidence associated with consumption of areca nut. Reduction or preferably stoppage of the habit forms an essential component of the total treatment plan. The mainstay in the treatment of OSMF is therefore concentrated upon improving mouth opening and relieving the symptoms either by medicinal or surgical means. The medicinal treatment for mild cases of OSMF includes steroids, cardiovascular drugs, antioxidants, vitamins and iron supplements. Topical application of steroids, hyaluronidase, collagenase, and placental extract has yielded positive results in mild cases but in advanced cases, surgery followed by aggressive physiotherapy is the only viable treatment which produces satisfactory results.

Excision of the fibrous bands and propping the mouth open to allow secondary epithelialisation causes rebound fibrosis during healing. Release of fibrous bands and split thickness skin grafting has a high recurrence from contracture. The survival of full thickness skin grafts is questionable. The use of island palatal flaps based on the greater palatine artery as recommended by Khanna et al. has limitations including involvement of the donor site by fibrosis, limited donor tissue with limited reach of the flap, and the need for extraction of maxillary second molars to cover the defect with the flap under no tension. The bilateral tongue flaps cause severe dysphasia, disarticulation, and carry the risk of postoperative aspiration. They also provide a limited amount of donor tissue as their reach is inadequate. The stability of a tongue flap and dehiscence are the common postoperative complications of uncontrolled tongue movements. Apart from this the reported involvement of the tongue is 38%, which precludes its use for reconstruction. Buccal fat pads may also be used to cover the defects after excision of the fibrous bands. The harvesting of the buccal fat pad is simple because access is easy. However, severe atrophy of buccal fat pads is seen in patients with chronic disease. In addition, the anterior reach of the buccal fat pad is often inadequate, and the region anterior to the cuspid is required to be left raw. This raw area heals by secondary intention and subsequently fibrosis, leading to gradual relapse. Bilateral radial forearm free flaps are hairy, 40% of patients require secondary debulking procedures, and the facilities for free tissue transfer are not universally available. Canniff and Harvey recommended temporal myotomy or coronoidectomy to release severe trismus caused by the atrophic changes in the tendon of temporalis muscle secondary to the disease.

The use of the nasolabial flap in reconstruction of head and neck defects has proved to be efficacious and reliable. The versatility of this flap has been attributed to the fact that there is often abundant non - hair bearing skin in this well vascularized region. Also the proximity to the defect and achievement of good cosmetic result with preservation of function and least distortion of anatomy makes it the flap of choice. Therefore, these advantages of 'extended single stage nasolabial flap' in the treatment of OSMF led us to carry out this study for "Evaluation of change in mouth opening in centimeters in oral submucous fibrosis patients after surgical excision of fibrous bands along with bilateral coronoidotomy & surgical defect coverage by single stage nasolabial flap". Mouth opening in centimeters was recorded pre operatively(base line),to 1 week,2 week,3 week,4 week, 2nd month,3rd month and 6 month post operatively and the change was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cases of OSMF based on thorough clinical examination and long standing positive history of habits such as chewing betel nut etc.
* Decreased mouth opening (less or equal to 25mm interincisal distance).
* Patients willing to quit habit.
* Intra orally palpable fibrous bands.

Exclusion Criteria:

* Mouth opening > 25 mm.
* Patients showing malignant changes in histopathological report.
* Medically compromised patients unfit for surgery under general anesthesia.
* Patients not willing to quit habit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Mouth opening in centimeters | Baseline
  comparison of pre operative,intra operative,1 week post operative , 2nd week, 3rd week,4th week, 2nd month,3rd month, 6th month post operative mouth opening.
Mouth opening in centimeters | 1week
Mouth opening in centimeters | 2week
Mouth opening in centimeters | 3week
Mouth opening in centimeters | 4 week
Mouth opening in centimeters | 2 month
Mouth opening in centimeters | 3 month
Mouth opening in centimeters | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: faisal idrees, mds, Principal Investigator — Government College of Dentistry, Indore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lazaridis N. Unilateral subcutaneous pedicled nasolabial island flap for anterior mouth floor reconstruction. J Oral Maxillofac Surg. 2003 Feb;61(2):182-90. doi: 10.1053/joms.2003.50045. PMID 12618994
- [Background] Yousif NJ, Gosain A, Matloub HS, Sanger JR, Madiedo G, Larson DL. The nasolabial fold: an anatomic and histologic reappraisal. Plast Reconstr Surg. 1994 Jan;93(1):60-9. PMID 8278485